CLINICAL TRIAL: NCT04813367
Title: Long Term Follow-up of Twisted Fallopian Tubes Among Young Girl. International Study
Brief Title: Twisted Fallopian Tubes
Acronym: Tubes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_0239
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Twisted Fallopian Tube
Keywords: Twisted Fallopian Tube

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Twisted fallopian tubes cohort: Description of girls who went through surgery for twisted fallopian tubes
  Interventions: Procedure: Surgery of twisted fallopian tubes

INTERVENTIONS:
Procedure: Surgery of twisted fallopian tubes — Patients diagnosed with twisted fallopian tube go through surgery.

SUMMARY:
Isolated tubal torsion is a very rare event already in adults (1: 1.5 million women), it remains exceptional in children without being able to find a prevalence in the literature. The causes can be malformative or idiopathic, but even that remains unknown.

Because of the scarcity, surgical treatment is not standardized and left to the good care of the surgeon in charge.

ELIGIBILITY:
Inclusion Criteria:

* Patient younger then 18 going through surgery for twisted fallopian tubes

Exclusion Criteria:

* Girl above 18 and tubal torsion associated with ovary torsion

Max Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Girl younger than 18 with isolated tubal torsion. Girl above 18 and tubal torsion associated with ovary torsion are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Fallopian tube Surgery results | Evaluation 10 years after surgery
  Evaluation of twisted fallopian surgery interest on then long terms, define as percentage of patients going through surgical revision

CONTACTS AND LOCATIONS:
Locations (13):
- France (4):
  - CHU Amiens, Amiens
  - Centre Hospitalier Universitaire de Angers, Angers
  - APHM, Hôpital La Timone Enfants et Hôpital Nord, Marseille
  - Hopital NECKER Enfant Malades, Paris
- Italy (6):
  - ASP Trapani - presidio ospedaliero "S. Antonio Abate, Erice
  - Azienda Ospedaliera Universitaria di Padova, Padua
  - AOU Siena, Ospedale le Scotte, Siena
  - Ospedale infantile Regina Margherita, Torino
  - Institute for Maternal and Child Health - IRCCS "Burlo Garofolo, Trieste
  - Institute for Maternal and Child Health IRCCS G. Gaslini, Genova, Trieste
- Hôtel-Dieu de France Hospital, Beirut, Lebanon
- Hospital d Urgences pour les enfants, Iași, Romania
- Ege University Faculty of Medicine Children's Hospital, Izmir, Turkey (Türkiye)